CLINICAL TRIAL: NCT01200797
Title: A Phase II Evaluation of SJG-136 in Women With Cisplatin-Refractory or Resistant Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Carcinoma
Brief Title: SJG-136 in Treating Patients With Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer That Did Not Respond to Previous Treatment With Cisplatin or Carboplatin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual was the reason for study termination.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02519; NCI-2011-02519 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-VICC-GYN-1003; CDR0000682791; VICC GYN 1003 (Other: H. Lee Moffitt Cancer Center and Research Institute); 8489 (Other: CTEP); N01CM00100 (NIH); NCT01199796 (obsolete NCT alias)
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — 1,1'-((propane-1,3-diyl)dioxy)bis(7-methoxy-2-methylidene-1,2,3,10,11,11a-hexahydro-5H-pyrrolo(2,1-c)(1,4)benzodiazepin-5,11-dione)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (SJG-136) (Experimental): Patients receive SJG-136 IV over 20 minutes on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: SJG-136; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: SJG-136 — Given IV
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well SJG-126 works in treating patients with epithelial ovarian, primary peritoneal, or fallopian tube cancer that did not respond to previous treatment with cisplatin or carboplatin. Drugs used in chemotherapy, such as SJG-136, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall response rate to SJG-136 in patients with persistent or recurrent platinum-refractory epithelial ovarian, primary peritoneal, or fallopian tube carcinoma.

II. To assess the nature and degree of toxicity of this regimen in these patients.

III. To determine other parameters of response, including progression-free survival, overall survival, and time to progression in patients treated with this regimen.

Correlative Endpoints:

I. To correlate response rates with the degree of DNA adduct formation in peripheral blood mononuclear cells (PBMCs) and tumor cells as measured by the single-cell gel electrophoresis (Comet) assay and γ-H2AX assay.

II. To assess whether the rate of DNA adduct formation in PBMCs correlates with the rate of DNA adduct formation in tumor cells.

III. To evaluate BRCA1 protein expression in archival tissue specimens from the patient's primary tumor reductive surgery.

IV. To determine the ability of BRCA1 protein in repairing/removing DNA-adducts in PBMCs and tumor tissue.

VI. To evaluate the effect of BRCA1 protein expression on the overall response rate to SJG-136.

OUTLINE: This is a multicenter study.

Patients receive SJG-136 IV over 20 minutes on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection at baseline and periodically during study for correlative studies. Tumor tissue samples may also be collected.

After completion of study therapy, patients are followed up for 30 days and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Must have persistent or recurrent epithelial ovarian, primary peritoneal, or fallopian tube carcinoma, with histologic confirmation of the original primary tumor.
* Must have had at least one prior platinum-based (cisplatin or carboplatin) chemotherapy regimen for the management of their primary disease. This would include intraperitoneal chemotherapy.
* Must be considered platinum refractory or resistant, defined as patients with progression of disease during platinum-based chemotherapy, patients having persistent disease at the completion of platinum-based chemotherapy, or patients having a disease free interval following prior platinum therapy of less than six months.
* May have had no more than three prior treatment regimens for their epithelial ovarian, primary peritoneal or fallopian tube carcinoma. Consolidation or maintenance therapy initiated within six weeks of the completion of primary therapy will not be counted as an additional regimen.
* Must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Time interval from last chemotherapy, radiotherapy, or surgery of at least four weeks and the patient must have recovered from any significant adverse effects of prior treatment. Patients must be at least six weeks from having received nitrosoureas or mitomycin C.
* Life expectancy greater than three months.
* Must have adequate bone marrow and organ function:

  * Leukocyte count > 3 x 10^9/L
  * Absolute neutrophil count (ANC) > 1.5 x 10^9/L
  * Platelet count > 100 x 10^9/L
  * Total bilirubin Within normal institutional limits
  * Aspartate aminotransferase (AST)/alanine transaminase (ALT) < 2.5 x institutional upper limits of normal
  * Creatinine < 1.5 mg/dL or calculated creatinine clearance (ClCr) > 60 ml/min by Cockcroft Gault method, as below. ClCr = weight (kg) x (140-age) x 0.85 72 x serum creatinine (mg/dL)
* Participants must have signed an approved informed consent.
* Participants of childbearing potential must have a negative serum pregnancy test prior to study entry and must use an effective form of contraception.
* Must have archival tissue available from their original tumor debulking surgery for assessment of BRCA1 protein expression.

Exclusion Criteria:

* Patients with borderline ovarian tumors, ovarian germ cell tumors, ovarian sex-cord stromal tumors, or other non-epithelial ovarian tumors are not eligible.
* Patients receiving any other investigational agents.
* Patients who have received radiation therapy to more than 25% of the bone marrow.
* Patients who have previously received SJG-136 or related compounds.
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with the study requirements.
* Prior malignancy (other than cervical carcinoma in situ, ductal carcinoma in situ of the breast, or non-melanoma skin cancer) unless treated with curative intent and without evidence of disease for three years.
* With the exception of alopecia (or other situations in which the organ dysfunction or symptoms are considered clinically insignificant or irrelevant to the study), patients may not have baseline organ dysfunction or symptoms that qualify as grade 2 or higher by the CTEP Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0. Particular attention should be paid to assessment of pre-existing edema, since vascular leak syndrome was the dose limiting toxicity of this agent in the phase I trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Crispens, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (6):
- United States (6):
  - Hartford Hospital, Hartford, Connecticut
  - Oncology Associates PC, Hartford, Connecticut
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual in July 2010, with participants enrolled from 11/1/2010 through 8/30/2012. Five Southeast Phase 2 Consortium (SEP2C) cancer center sites participated in this study.
Pre-assignment Details: Twenty-two patients consented to this study. Three were not eligible to receive treatment.
Groups:
- Treatment (SJG-136): SJG-136 was administered consecutively on days 1 - 3 as a 20-minute intravenous infusion, at a dose of 30 mcg/m2/day. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (SJG-136)
Started | 19
Completed | 0
Not Completed | 19
Not completed — symptomatic deterioration | 2
Not completed — Adverse Event | 4
Not completed — Disease Progression | 13

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Treatment (SJG-136)
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 60.57895 [35 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR)
Description: Number of patients in each response category, per RECIST v1.1, summarized as follows for target lesion criteria (see RECIST v1.1 for additional details): complete response (CR),disappearance of target lesions; partial response (PR), >=30% decrease in sum of longest diameter (LD) of target lesions; progressive disease (PD), >=20% increase in sum of LD of target lesions or appearance of new lesions; stable disease (SD), insufficient change in target lesions or new lesions to qualify as either PD or PR. Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>SD>PD. Confirmation of CR or PR is required to deem either one the best overall response.
Time Frame: On-treatment date to date of disease progression (assessed up to 12 months)
Population: All patients with best overall response data; patients are excluded if best overall response data is missing or if the patient is nonevaluable for best overall response
Measure: Number; unit: participants
Groups:
- Treatment (SJG-136): Patients receive 30 mcg/m2 of SJG-136 intravenously, over a period of 20 minutes, on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (SJG-136)
Number analyzed (Participants) | 17
participants
  Number of patients with complete response | 0
  Number of patients with partial response | 0
  Number of patients with stable disease | 6
  Number of patients with progressive disease | 11
  Number of patients not evaluable | 2

2. Primary Outcome: Number of Patients With Each Worst-grade Toxicity
Description: Count of patients according to the worst-grade toxicity experienced by each, where worst-grade toxicity is per NCI common toxicity criteria: grade 1, mild; grade 2, moderate; grade 3, severe; grade 4, life-threatening; grade 5, death.
Time Frame: On-study date to 30 days following final dose of study
Population: Total number of patients reported with any toxicity. Not all participants may have an adverse event, thus not every patient on-treatment may be accounted for in worst-grade toxicities.
Measure: Number; unit: participants
Groups:
- Treatment (SJG-136): Patients receive 30 mcg/m2 of SJG-136 intravenously, over a period of 20 minutes, consecutively on days 1-3. Treatment courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (SJG-136)
Number analyzed (Participants) | 18
participants
  Number of patients with worst-grade toxicity 1 | 5
  Number of patients with worst-grade toxicity 2 | 8
  Number of patients with worst-grade toxicity 3 | 4
  Number of patients with worst-grade toxicity 4 | 1
  Number of patients with worst-grade toxicity 5 | 0

3. Primary Outcome: Progression-free Survival (PFS)
Description: Estimated probable duration of life without disease progression, from on-study date to earlier of progression date or date of death from any cause, using the Kaplan-Meier method with censoring (see analysis population description for additional details). Disease progression is defined under RECIST v1.1 as >=20% increase in sum of longest diameters of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Time Frame: On-study date to lesser of date of progression or date of (assessed up to 12 months)
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where either death or progression is an event, with censoring for non-progressed, non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (SJG-136)
Number analyzed (Participants) | 19
days | 49 [44 to 79]

4. Primary Outcome: Overall Survival (OS)
Description: Estimated probable duration of life from on-study date to date of death from any cause, using the Kaplan-Meier method with censoring (see analysis population description for additional details).
Time Frame: On-study date to date of death from any cause (assessed up to 12 months)
Population: All patients are included in the analysis on intention-to treat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: daya
Arm/Group | Treatment (SJG-136)
Number analyzed (Participants) | 19
daya | 271 [145 to 371]

5. Primary Outcome: Time to Progression (TTP)
Description: Estimated probable duration from on-study date to date of disease progression, using the Kaplan-Meier method with censoring (see analysis population description for additional details). Disease progression is defined under RECIST v1.1 as >=20% increase in sum of longest diameters of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Time Frame: On-study date to date of progression (assessed up to 12 months)
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where progression is an event, with censoring for non-progressed patients at greater of off-study date, last known alive date, or date of death not attributable to disease progression.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (SJG-136)
Number analyzed (Participants) | 19
days | 49 [44 to 129]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment (SJG-136)
Serious Adverse Events (participants affected / at risk) | 9/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SJG-136) (N=19)
Heart failure (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain - Grade 2 (Gastrointestinal disorders) | 2 (2)
Abdominal pain - Grade 3 (Gastrointestinal disorders) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea - Grade 2 (Gastrointestinal disorders) | 1 (1)
Nausea - Grade 3 (Gastrointestinal disorders) | 2 (2)
Vomiting - Grade 1 (Gastrointestinal disorders) | 1 (2)
Vomiting - Grade 2 (Gastrointestinal disorders) | 1 (1)
Vomiting - Grade 3 (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Edema trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
General disorders and administration site conditions - other (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Injury - other (car crash) (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Dyspnea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SJG-136) (N=19)
Fatigue (General disorders) | 9 (11)
Edema limbs (General disorders) | 7 (8)
Pain (General disorders) | 3 (5)
General disorders and administration site conditions - other (General disorders) | 2 (2)
Edema face (General disorders) | 1 (1)
Edema trunk (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (10)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Metabolism and nutrition disorders - other (Metabolism and nutrition disorders) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (12)
Vomiting (Gastrointestinal disorders) | 8 (11)
Constipation (Gastrointestinal disorders) | 7 (9)
Abdominal pain (Gastrointestinal disorders) | 6 (9)
Ascites (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Weight gain (Investigations) | 5 (7)
Lymphocyte count decreased (Investigations) | 4 (7)
Alkaline phosphatase increased (Investigations) | 2 (3)
Creatinine increased (Investigations) | 2 (2)
Investigations - other (Investigations) | 1 (2)
Lymphocyte count increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - other (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (10)
Blood and lymphatic system disorders - other (Blood and lymphatic system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorders - other (Nervous system disorders) | 1 (2)
Parethesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (2)
Phlebitis (Vascular disorders) | 1 (2)
Vascular disorders - other (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1)
Renal and urinary disorders - other (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Eye disorders - other (Eye disorders) | 1 (1)
Neoplasms benigh, malignant and unspecified (incl cysts and polyps) - other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The death reported in the SAE section was not related to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less